CLINICAL TRIAL: NCT05474768
Title: Expectations and Beliefs of Transgender People Regarding Hormonal Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, EVA FEIGERLOVA, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI221
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Transgenderism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Hormonal treatment of gender dysphoria can have repercussions on metabolism, cardiovascular system and fertility and represents à potential oncological risk. According to the recommendations of the Endocrine society. Therefore, initial assessment and follow-up visits are necessary and must be carried out to avoid the apparition of potentially undesirable effects.

ELIGIBILITY:
Inclusion Criteria:

* being a parent of adolescent/child presenting Gender dysphoria
* adult subject (age > 18 years) presenting Gender dysphoria

non-inclusion criteria

* Severe, uncontrolled psychiatric or somatic illness
* Chronic alcoholism
* Substance abuse
* Refusal or linguistic, physical or psychological incapacity to participate in the study
* Ongoing pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with gender dysphoria and parent of adolescent/child presenting gender dysphoria, who are followed un the university hospital of Nancy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Describe expectations and beliefs of transgener people about hormonal therapy | 12 months
  qualitative analysis of qualitative data from collective discussions (focus groups)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France